CLINICAL TRIAL: NCT00661531
Title: A Single Arm Phase II Study of Pharmacologic Dose Estrogen in Postmenopausal Women With Hormone Receptor-Positive Metastatic Breast Cancer After Failure of Sequential Endocrine Therapies
Brief Title: Estrogen in Postmenopausal Women With ER Positive Metastatic Breast Cancer After Failure of Sequential Endocrine Therapy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Poor accrual
Sponsor: Georgetown University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FER-BR-030; W81XWH-06-1-0590 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2008-04-17; First posted 2008-04-18 (Estimated); Results first posted 2017-03-07 (Actual); Last update posted 2017-04-12 (Actual); Status verified 2015-11

CONDITIONS: Breast Cancer; Cancer of the Breast; Neoplasms, Breast
Keywords: Breast cancer; Metastatic breast cancer; ER positive breast cancer; Hormonal therapy
MeSH Terms: conditions — Breast Neoplasms | interventions — Estradiol; Anastrozole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Estrace & Anastrozole (Experimental): Estrace 10 mg three times a day for 3 months. After 3 months of estrace, the estrace will be stopped and anastrazole 1 mg daily will be administered
  Interventions: Drug: Estrace; Drug: Anastrozole

INTERVENTIONS:
Drug: Estrace — Estrace 10 mg three times daily will be administered for 3 months.
Drug: Anastrozole — After 3 months of estrace, patients who do not have evidence of disease progression will then be switched to received Anastrozole 1 mg daily as long as their disease benefits from this treatment
  Other Names: Arimidex

SUMMARY:
This trial seeks to confirm the response rate for estrace treatment in a patients with hormone receptor positive metastatic breast cancer heavily pre-treated with modern endocrine therapies.

DETAILED DESCRIPTION:
Prior to the current standard of care utilizing estrogen deprivation or antiestrogen therapy to treat hormonally sensitive breast cancers, treatment with pharmacologic doses of estrogen was a common technique used to treat post-menopausal women with hormone sensitive metastatic disease that resulted in durable responses with regression of disease. A randomized trial comparing tamoxifen and pharmacologic doses of estrogen demonstrated similar rates of response with long-term follow-up data confirming a survival benefit for those treated with the estrogen preparation. Additional data has shown that post-menopausal women with hormonally sensitive tumors that have progressed on prior endocrine therapies responded to treatment with pharmacologic doses of estrogen. These data, coupled with pre-clinical data that postmenopausal levels of estrogen can be used to cause apoptosis (programmed cell death within the tumor) and tumor regression in exhaustively treated endocrine resistant disease form the rationale for the proposed clinical trial. This trial seeks to confirm the response rate for estrace treatment in a patient population heavily pre-treated with modern endocrine therapies.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed estrogen and/or progesterone receptor-positive breast cancer metastatic breast cancer
* Clinically determined evaluable disease
* Post-menopausal woman
* Previous clinical benefit from prior anti-estrogen therapies and subsequent failure of at least 2 prior endocrine therapies.
* May have had chemotherapy for adjuvant &/or metastatic disease.
* May have had radiation therapy but not to the only site of disease.
* Ecog performance status </= 2.
* Life expectancy of > 6 months

Exclusion Criteria:

* Chemotherapy or radiotherapy within 1 week of beginning treatment in the clinical trial
* Brain metastasis
* Prior history of or active thrombophlebitis, deep venous thrombosis or pulmonary embolus
* Current vaginal bleeding
* Hypercalcemia or hypocalcemia
* History of or active hepatic adenoma
* No other malignancies within the past 5 years with the exception of curatively treated basal cell or squamous cell carcinoma of the skin or carcinoma in-situ of the cervix

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2008-04; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Claudine Isaacs, M.D., Principal Investigator — Lombardi Comprehensive Cancer Center
Locations (3):
- United States (3):
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - Cooper Cancer Institute, Voorhees Township, New Jersey
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Estrace & Anastrozole
Started | 11
Completed | 8
Not Completed | 3
Not completed — Withdrawal by Subject | 3

BASELINE CHARACTERISTICS:
Arm/Group | Estrace & Anastrozole
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 4
Age, Continuous [Median (Full Range); unit: years] | 64 [53 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 10
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 11

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival
Description: Progression free survival is defined as the time from assignment of treatment to the time of disease progression or death from any cause
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Estrace & Anastrozole
Number analyzed (Participants) | 11
Participants | 7

2. Secondary Outcome: Response Rate
Description: Response rate was defined per RECIST version 1.0. In this study, response rate was defined as including patients with either a complete response (complete disappearance of all target lesions with changes confirmed by repeat assessments performed no less than 4 weeks after the criteria for response was first met) or a partial response (at least 30% decrease in the sum of the longest diameter of the target lesions)
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Estrace & Anastrozole
Number analyzed (Participants) | 11
Participants | 2

ADVERSE EVENTS:
Arm/Group | Estrace & Anastrozole
Serious Adverse Events (participants affected / at risk) | 2/11
Other Adverse Events (participants affected / at risk) | 11/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Estrace & Anastrozole (N=11)
Anal Hemorrhage (Gastrointestinal disorders) | 1 (1) — Hemorrhoidal bleed with hypotension requiring admission - treated with intravenous fluids and correction of INR
Hypercalcemia (Metabolism and nutrition disorders) | 1 (11) — Admitted with confusion, nausea, and mental status change. Found to haver hypercalcemia and treated with hydration
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Estrace & Anastrozole (N=11)
Anemia (Blood and lymphatic system disorders) | 6 (11)
Rhinitis (Infections and infestations) | 4 (7)
Neutropenia (Blood and lymphatic system disorders) | 1 (1)
Lymphopenia (Blood and lymphatic system disorders) | 7 (9)
Lymphedema (Vascular disorders) | 2 (3)
Edema (Vascular disorders) | 4 (5)
Hypertension (Cardiac disorders) | 2 (5)
Hot flashes (Vascular disorders) | 3 (3)
Dizziness (Nervous system disorders) | 4 (4)
Fatigue (General disorders) | 9 (12)
Anxiety (Psychiatric disorders) | 2 (2)
Chills (General disorders) | 3 (3)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (4)
Vaginal bleeding (Reproductive system and breast disorders) | 6 (7)
Rash (Skin and subcutaneous tissue disorders) | 1 (4)
Nausea (Gastrointestinal disorders) | 8 (10)
Emesis (Gastrointestinal disorders) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 3 (3)
Constipation (Gastrointestinal disorders) | 4 (5)
Anorexia (Gastrointestinal disorders) | 4 (5)
Insomnia (Psychiatric disorders) | 4 (5)
Depression (Psychiatric disorders) | 2 (2)
Neuropathy (Nervous system disorders) | 2 (4)
Abdominal pain (Gastrointestinal disorders) | 3 (3)
Bone pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Weakness generalized (Musculoskeletal and connective tissue disorders) | 4 (5)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4 (11)
Breast pain (Reproductive system and breast disorders) | 6 (7)
Headache (Nervous system disorders) | 4 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (14)
Dypsnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 7 (12)
Aspartate aminotransferase elevation (Investigations) | 5 (5)
Alkaline phosphotase elevation (Investigations) | 7 (15)
Alanine aminotransferase elevation (Investigations) | 4 (7)
Hyperglycemia (Metabolism and nutrition disorders) | 9 (21)
Hypercalcemia (Metabolism and nutrition disorders) | 3 (3)
Hypocalcemia (Metabolism and nutrition disorders) | 2 (6)
Infection (Infections and infestations) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No